CLINICAL TRIAL: NCT07269301
Title: A PHASE 1, OPEN-LABEL, SINGLE-DOSE, PARALLEL-COHORT STUDY TO EVALUATE THE PHARMACOKINETICS, SAFETY, AND TOLERABILITY OF PF-07328948 IN ADULTS WITH AND WITHOUT VARYING DEGREES OF HEPATIC IMPAIRMENT
Brief Title: A Study to Learn How the Body Processes the Study Medicine PF-07328948 in People With and Without Reduced Liver Function
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C4921011; C4921011 (Other: Pfizer)
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Hepatic Impairment; Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1: PF-07328948 participants with severe hepatic impairment (Experimental): Participants with severe hepatic impairment will receive a single dose of PF-07328948, administered orally as 1 PF-07328948 tablet.
  Interventions: Drug: PF-07328948
- Group 2: PF-07328948 participants with moderate hepatic impairment (Experimental): Participants with moderate hepatic impairment will receive a single dose of PF-07328948, administered orally as 1 PF-07328948 tablet.
  Interventions: Drug: PF-07328948
- Group 3: PF-07328948 participants with mild hepatic impairment (Experimental): Participants with mild hepatic impairment will receive a single dose of PF-07328948, administered orally as 1 PF-07328948 tablet.
  Interventions: Drug: PF-07328948
- Group 4: PF-07328948 participants without hepatic impairment (Experimental): Participants without hepatic impairment will receive a single dose of PF-07328948, administered orally as 1 PF-07328948 tablet.
  Interventions: Drug: PF-07328948

INTERVENTIONS:
Drug: PF-07328948 — PF-07328948, 1 tablet orally, once on Day 1

SUMMARY:
The purpose of this study is to understand the effects of decreased liver function on the study medicine (PF-07328948). People with decreased liver function may process the study medicine differently from healthy people.

Study is seeking participants who:

* Are between 18 and 75 years of age.
* Have a BMI (body mass index) of 17.5 to 40 kg/m2, inclusive, and a total body weight of more than or equal to 45 kilograms or 99 pounds.

Participants will take the study medicine as a tablet once at the study clinic and then will stay onsite for about 6 days.

During this time, the study team will check for the participant's treatment experience and take some blood samples to test the level of PF-07328948. This will help understand if certain level of decreased liver function could affect the study medicine being processed in the body.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of nonchildbearing potential, between the ages of 18 (inclusive) and 75 years, at the screening visit.
* Willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
* BMI of 17.5 to 40.0 kg/m2 (inclusive), and a total body weight ≥45 kg (99 lb).
* Group 4 only: at screening, no clinically relevant abnormalities identified by a detailed medical history, physical exam, including blood pressure and pulse rate measurement, ECG and clinical laboratory tests.
* Group 4 only: no known or suspected hepatic impairment and meet the criteria based on screening laboratory liver function tests.
* Groups 1, 2 & 3 only: stable hepatic impairment that meets criteria for Class A, B, or C of the Child-Pugh classification with no clinically significant change in disease status within 28 days before screening.
* Groups 1, 2 & 3 only: stable concomitant medications for the management of individual participant's medical history.

Exclusion Criteria:

* Any condition possibly affecting drug absorption
* At screening, a positive result for HIV antibodies.
* Evidence of a prothrombotic state, including history of deep vein thrombosis, pulmonary embolism, or arterial thrombosis, or known genetic predisposition.
* Other medical or psychiatric condition or laboratory abnormality that may increase the risk of study participation or make the participant inappropriate for the study.
* Use of specific prohibited prior/concomitant therapies
* Use of an investigational product within 30 days or 5 half-lives (whichever longer).
* eGFR<60 mL/min/1.73m2 at screening.
* A positive urine drug test at screening or admission to study clinic.
* At screening or admission to study clinic, a positive breath alcohol test.
* History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of screening.
* Group 4 only: evidence of chronic liver disease including history of hepatitis, hepatitis B, or hepatitis C.
* Group 4 only: screening ECG demonstrating QTcF interval >450 ms or a QRS interval >120 ms.
* Group 4 only: screening seated systolic blood pressure ≥140 mm Hg or diastolic blood pressure ≥90 mm Hg
* Group 1, 2 & 3 only: Hepatic carcinoma or hepatorenal syndrome or limited predicted life expectancy (defined as <1 year in Groups 2 & 3 and <6 months for Group 1 only).
* Group 1, 2 & 3 only: a diagnosis of hepatic dysfunction secondary to any acute ongoing hepatocellular process that is documented by medical history, physical exam, liver biopsy, hepatic ultrasound, CT scan, or MRI.
* Group 1, 2 & 3 only: history of gastrointestinal hemorrhage due to esophageal varices or peptic ulcers less than 4 weeks prior to screening.
* Group 1, 2 & 3 only: signs of clinically active Grade 3 or 4 hepatic encephalopathy
* Groups 1, 2 & 3 only: severe ascites and/or pleural effusion, except for those categorized in Group 4 who may be enrolled provided participant is medically stable, per the study doctor's judgment.
* Groups 1, 2 & 3 only: previously received a kidney, liver, or heart transplant.
* Groups 1, 2, & 3 only: screening ECG demonstrating a QTcF interval >470 ms or a QRS interval >120 ms.
* Groups 1, 2 & 3 only: persistent severe, uncontrolled hypertension at screening, admission to study clinic, or pre-dose on Day 1.
* Groups 1, 2 & 3 only: ALT or AST >5x upper limit of normal on clinical laboratory tests at screening.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-12-22 (Actual); Primary Completion 2027-02-23 (Estimated); Study Completion 2027-02-23 (Estimated)

PRIMARY OUTCOMES:
Fraction of Unbound Drug in Plasma (Fu) of PF-07328948 | At 0 (prior to dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, and 168 hours post dose on Day 1
  Fu is the fraction of unbound drug in plasma, which is calculated by Cu/C (where Cu represents unbound concentration and C represents total concentration).
Unbound AUCinf (AUCinf,u) of PF-07328948 | At 0 (prior to dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, and 168 hours post dose on Day 1
  AUCinf is the area under the plasma concentration-time profile from time zero extrapolated to infinite time. AUCinf,u is the unbound AUCinf.
Unbound Cmax (Cmax,u) of PF-07328948 | At 0 (prior to dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, and 168 hours post dose on Day 1
  Cmax is the maximum plasma concentration. Cmax,u is the unbound Cmax.

SECONDARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (TEAEs) | Day 1 to Day 36

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - Orange County Research Center, Lake Forest, California
  - Orlando Clinical Research Center, Orlando, Florida
  - Genesis Clinical Research, LLC, Tampa, Florida

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4921011